CLINICAL TRIAL: NCT02831439
Title: A Statewide Intervention to Reduce Use of Unproven or Ineffective Breast Cancer Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Collaborators: Wisconsin Collaborative for Healthcare Quality (Unknown); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Ann Nattinger, Senior Associate Dean for Research, Lady Riders Professor of Breast Cancer Research, Professor of Medicine, Medical College of Wisconsin
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: PRO00022912; R01CA190016 (NIH)
Record Dates: First submitted 2016-06-21; First posted 2016-07-13 (Estimated); Last update posted 2020-01-22 (Actual); Status verified 2020-01

CONDITIONS: Breast Cancer
Keywords: Choosing Wisely; Breast cancer; Controlled trial; High-value health care; Health services research
MeSH Terms: conditions — Breast Neoplasms | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Participating health systems in Wisconsin. Interventions include: Basic public reporting and the enhanced intervention (app)
  Interventions: Behavioral: Basic public reporting; Behavioral: Enhanced intervention
- Control (Other): Health systems in comparison states. Control includes: Cost savings comparison
  Interventions: Behavioral: Control group - observational

INTERVENTIONS:
Behavioral: Basic public reporting — The basic intervention will comprise public reporting through the WCHQ website. Individual-level, claims data submitted for billing to third party payers by participating healthsystems will be used to (i) identify cohorts of women with incident breast cancer at the practice-level and (ii) construct the metrics for public reporting and individual benchmarking information. These data are consistent with Medicare and Marketscan claims in both format and content thereby ensuring seamless application of the validated algorithm as well as construction of outcome variables as proposed in Aims 1 and 2 of the study.
  Arms: Intervention
Behavioral: Enhanced intervention — The enhanced intervention adds an app comprising a decision tool, patient education and communication information that will be delivering concise, readily accessible information about the main components of the intervention. Specifically, physicians in participating practices will be provided a smartphone-based, point-of-care application that will include i) a list of the unproven/ineffective interventions with statements about a) scientifically proven appropriate use; b) proven or suspected downsides to inappropriate use; ii) clinical calculators that allow physician to input individual patients' clinical/tumor characteristics for each test; iii) practice-specific summary of publicly reported results; and iv) printable patient information adapted from the ASCO Choosing Wisely website.
  Arms: Intervention
Behavioral: Control group - observational — Comparison states will be used to evaluate the interventions in light of possible secular trends in the region and the nation. The design strategy will enable estimates of the effectiveness of the basic intervention (Aim 1) by comparing (i) the pre-intervention rates to post-intervention rates as well as by comparing (ii) changes between the pre- and post-intervention periods for the "treatment" state (WI) relative to comparison states, neighboring states and others. A similar approach will be used in Part II to provide estimates of the enhanced intervention's impact relative to the basic intervention and contemporary usual care provided in control states, thereby enabling the cost-savings analyses proposed as part of Aim 3.
  Other Names: Control group
  Arms: Control

SUMMARY:
The goal of this project is to examine the effectiveness and potential cost savings of two organizational interventions aimed at reducing the use of ineffective or unproven care among women with incident breast cancer.

DETAILED DESCRIPTION:
Challenged by public opinion, peers and the Congressional Budget Office, a number of specialty societies have recently begun to develop "Top Five" lists of relatively expensive procedures that do not provide meaningful benefit to at least some categories of patients for whom they are commonly ordered. The Choosing Wisely® campaign is the most visible example. The extent to which the development of these lists has influenced the behavior of physicians or patients, however, remains unknown.

In this study, investigators partner with the Wisconsin Collaborative for Healthcare Quality (WCHQ), a statewide consortium of hospitals, medical practices and health systems, to examine the effectiveness of two organizational interventions in reducing unproven or ineffective breast cancer care. Two interventions will be tested: (a) A "basic" public reporting intervention which summarizes on a public website practice-level statistics regarding use of targeted ineffective or unproven interventions for breast cancer and (ii) an "enhanced" intervention, augmenting public reporting with a smart phone-based application (App) that gives providers just-in-time information, decision-making tools, and personalized patient education materials that support reductions in the use of breast cancer interventions targeted based upon Choosing Wisely® or national oncology society guidelines. Specifically, the aims are: (1) To examine whether basic public reporting reduces use of targeted breast cancer practices among a contemporary cohort of patients with incident breast cancer in the intervention state relative to usual care in comparison states, using Marketscan and Medicare claims data while adjusting for possible confounders and temporal trends; (2) To examine the effectiveness of the enhanced intervention relative to the basic intervention; and (3) To simulate cost savings forthcoming from nationwide implementation of both interventions (relative to each other and to usual care) and to describe the implications of these findings for reimbursement policy and program initiatives.

The results will provide rigorous evidence regarding the effectiveness of a unique all-payer, all-age public reporting system for influencing provider behavior that may be easily exportable to other states. Findings will be further relevant to the ACO environment, which is expected to provide financial disincentives for providing ineffective or unproven care.

ELIGIBILITY:
Inclusion Criteria:

I. Health care providers: Health care providers (regardless of age, gender or race/ethnicity) in participating WCHQ practices who will provide breast cancer care to about 9,000 women who had an incident breast cancer surgery between 2014-2017.

II. Patients: Medicare and Marketscan women who had an incident breast cancer surgery between 2014-2017. No exclusions will be made by age or race/ethnicity. The focus on women is dictated by the very low prevalence of breast cancer among men.

Identification of incident breast cancer surgery in these datasets will be done using a validated algorithm developed by Nattinger et al.

Exclusion Criteria:

* Male patients are excluded from this analysis due to the low prevalence of breast cancer among males.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400415 (Actual)
Dates: Start 2014-09; Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Percentage of Women who received Intensity Modulated Radiation Therapy (IMRT) after Breast Conserving Surgery (defined as CPT 77418, 77385, 77386). | Date of surgery plus 180 days
  The American Society for Radiation Oncology's Choosing Wisely® list recommends against performing IMRT, a 3-dimensional technique that has not been demonstrated to provide a significant clinical advantage over the standard 2-dimensional technique for whole breast radiation therapy after breast conserving surgery.
Percent of Women had a CPM | Date of ipsilateral mastectomy surgery plus 1 day. Excluded from denominator if had any genetic predisposition counseling, testing, or family history codes within 180-days prior to surgery.
  (CPT 19303 OR 19304 w/mod 50; OR ICD-9 85.35 OR 85.36 OR 85.42; OR two claims within 1 day with ICD-9 85.33 OR 85.34 OR 85.41 OR 85.43 OR 85.45 OR 85.47, EXCLUDING two 85.45 OR two 85.47 OR (85.45 AND 85.47); OR conditions (a) AND (b) The National Comprehensive Cancer Network and the Society of Surgical Oncology indicate that there are no proven survival benefits to performing a Contralateral Prophylactic Mastectomy (CPM: removal of the unaffected breast). Despite the lack of survival benefit, this procedure may be considered appropriate in cases where there is high risk of cancer occurring in the unaffected breast and/or radiographic surveillance of the unaffected breast would be difficult. Such factors may include genetic predisposition to breast cancer, strong family history of breast cancer, high-risk histology (atypical hyperplasia or lobular carcinoma in situ), prior radiation treatment to the chest, and dense breast tissue.
Percentage of Women who received Tumor Biomarker Blood Testing for Surveillance (defined as CPT 82378 (CEA); 86300 (CA 15-3) | From 181 days post-date of surgery up to 4 years
  The American Society of Clinical Oncology's Choosing Wisely® list recommends against performing tumor biomarker blood tests (CA 15-3, CA 27.29, CEA) for breast cancer surveillance in asymptomatic women who have been treated with curative intent. Tumor markers may be indicated if there is concern for disease recurrence (development of symptoms or abnormal imaging findings).
Percentage of Women who received PET Scan or PET-CT Scan for Surveillance (defined as CPT 78811-78816; HCPCS G0235, G0252, S8085) | From 181 days post-date of surgery up to 4 years
  The American Society of Clinical Oncology's Choosing Wisely® list recommends against performing a positron emission tomography (PET) scan or a positron emission tomography-computed tomography (PET-CT) scan for routine breast cancer surveillance in asymptomatic patients who have been treated with curative intent, citing their unproven effectiveness in improving survival. PET/PET-CT scan may be indicated if there is concern for disease recurrence (development of symptoms or lab abnormalities) or to follow-up a prior abnormal PET/PET-CT scan finding.
Percentage of Women who received CT Scan for Surveillance (defined as CPT 71250, 71260, 71270, 72192-72194, 74150, 74160, 74170, 74176-74178) | From 181 days post-date of surgery up to 4 years
  The American Society of Clinical Oncology's Choosing Wisely® list recommends against performing a computerized tomography (CT or CAT) scan of the chest, abdomen or pelvis for routine breast cancer surveillance in asymptomatic patients who have been treated with curative intent, citing their unproven effectiveness in improving survival. CT scan may be indicated if there is concern for disease recurrence (development of symptoms or lab abnormalities) or to follow-up a prior abnormal CT scan finding.
Percentage of Women who received Bone Scan for Surveillance (defined as CPT 78306) | From 181 days post-date of surgery up to 4 years
  The American Society of Clinical Oncology's Choosing Wisely® list recommends against performing a bone scan for routine breast cancer surveillance in asymptomatic patients who have been treated with curative intent, citing their unproven effectiveness in improving survival. Bone scan may be indicated if there is concern for disease recurrence (development of symptoms or lab abnormalities) or to follow-up a prior abnormal bone scan finding.
Percentage of Women who received Breast MRI for Surveillance (defined as CPT 77058, 77059; HCPCS C8903-8908) | From 181 days post-date of surgery up to 4 years
  The American Society of Clinical Oncology, the American Cancer Society and the American Society of Breast Surgeons recommend against performing a breast magnetic resonance imaging (MRI) for routine breast cancer surveillance in asymptomatic patients who have been treated with curative intent, citing their unproven effectiveness in improving survival. Breast MRI is currently recommended only for women at very high risk for developing another breast cancer, such as BRCA1/2 mutation carriers, history of chest wall radiation therapy and women with a 20% or greater lifetime risk of developing another breast cancer. Breast MRI may be considered in patients with very dense breasts or a strong family history of breast cancer. Breast MRI may also be indicated for follow-up of a prior abnormal breast MRI finding.
Percentage of Women who received Follow-Up Mammograms More Frequently than Annually for Patients Treated with Breast Conserving Surgery & Radiotherapy (defined as CPT 77051, 77052, 77055-77057, 77061-77063 HCPCS G0202, G0204, G0206, G0279) | From 365 days post-surgery to 730 days post-surgery
  The American Society for Radiation Oncology's Choosing Wisely® list recommends against performing routine follow-up mammograms more frequently than annually in asymptomatic patients treated with breast conserving surgery and radiotherapy, citing no clear advantage to shorter interval imaging.

SECONDARY OUTCOMES:
Secondary costs associated with breast cancer care | From date of initial diagnosis up to 24 months
  Direct medical care costs for the initial diagnosis and evaluation, initial treatment as well as any neoadjuvant, adjuvant and surveillance care received during the first 24 months post-diagnosis will be calculated using Marketscan and Medicare claims data.

CONTACTS AND LOCATIONS:
Overall Officials: Ann Nattinger, MD, MPH, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Medical College of Wisconsin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yen TW, Laud PW, Sparapani RA, Nattinger AB. Surgeon specialization and use of sentinel lymph node biopsy for breast cancer. JAMA Surg. 2014 Feb;149(2):185-92. doi: 10.1001/jamasurg.2013.4350. PMID 24369337
- [Background] Grimshaw JM, Thomson MA. What have new efforts to change professional practice achieved? Cochrane Effective Practice and Organization of Care Group. J R Soc Med. 1998;91 Suppl 35(Suppl 35):20-5. doi: 10.1177/014107689809135S06. No abstract available. PMID 9797746
- [Background] Davis DA, Taylor-Vaisey A. Translating guidelines into practice. A systematic review of theoretic concepts, practical experience and research evidence in the adoption of clinical practice guidelines. CMAJ. 1997 Aug 15;157(4):408-16. PMID 9275952
- [Background] Bero LA, Grilli R, Grimshaw JM, Harvey E, Oxman AD, Thomson MA. Closing the gap between research and practice: an overview of systematic reviews of interventions to promote the implementation of research findings. The Cochrane Effective Practice and Organization of Care Review Group. BMJ. 1998 Aug 15;317(7156):465-8. doi: 10.1136/bmj.317.7156.465. No abstract available. PMID 9703533
- [Background] Grimshaw JM, Shirran L, Thomas R, Mowatt G, Fraser C, Bero L, Grilli R, Harvey E, Oxman A, O'Brien MA. Changing provider behavior: an overview of systematic reviews of interventions. Med Care. 2001 Aug;39(8 Suppl 2):II2-45. PMID 11583120
- [Background] Balas EA, Austin SM, Mitchell JA, Ewigman BG, Bopp KD, Brown GD. The clinical value of computerized information services. A review of 98 randomized clinical trials. Arch Fam Med. 1996 May;5(5):271-8. doi: 10.1001/archfami.5.5.271. PMID 8620266
- [Background] Chueh H, Barnett GO. "Just-in-time" clinical information. Acad Med. 1997 Jun;72(6):512-7. doi: 10.1097/00001888-199706000-00016. PMID 9200584
- [Background] Cabana MD, Rand CS, Powe NR, Wu AW, Wilson MH, Abboud PA, Rubin HR. Why don't physicians follow clinical practice guidelines? A framework for improvement. JAMA. 1999 Oct 20;282(15):1458-65. doi: 10.1001/jama.282.15.1458. PMID 10535437
- [Background] Davis DA, Thomson MA, Oxman AD, Haynes RB. Changing physician performance. A systematic review of the effect of continuing medical education strategies. JAMA. 1995 Sep 6;274(9):700-5. doi: 10.1001/jama.274.9.700. PMID 7650822
- [Background] Fung CH, Lim YW, Mattke S, Damberg C, Shekelle PG. Systematic review: the evidence that publishing patient care performance data improves quality of care. Ann Intern Med. 2008 Jan 15;148(2):111-23. doi: 10.7326/0003-4819-148-2-200801150-00006. PMID 18195336
- [Background] Ketelaar NA, Faber MJ, Flottorp S, Rygh LH, Deane KH, Eccles MP. Public release of performance data in changing the behaviour of healthcare consumers, professionals or organisations. Cochrane Database Syst Rev. 2011 Nov 9;(11):CD004538. doi: 10.1002/14651858.CD004538.pub2. PMID 22071813
- [Background] Berwick DM, James B, Coye MJ. Connections between quality measurement and improvement. Med Care. 2003 Jan;41(1 Suppl):I30-8. doi: 10.1097/00005650-200301001-00004. PMID 12544814
- [Background] Smith MA, Wright A, Queram C, Lamb GC. Public reporting helped drive quality improvement in outpatient diabetes care among Wisconsin physician groups. Health Aff (Millwood). 2012 Mar;31(3):570-7. doi: 10.1377/hlthaff.2011.0853. PMID 22392668
- [Background] Lamb GC, Smith MA, Weeks WB, Queram C. Publicly reported quality-of-care measures influenced Wisconsin physician groups to improve performance. Health Aff (Millwood). 2013 Mar;32(3):536-43. doi: 10.1377/hlthaff.2012.1275. PMID 23459733
- [Background] Mariotto AB, Yabroff KR, Shao Y, Feuer EJ, Brown ML. Projections of the cost of cancer care in the United States: 2010-2020. J Natl Cancer Inst. 2011 Jan 19;103(2):117-28. doi: 10.1093/jnci/djq495. Epub 2011 Jan 12. PMID 21228314
- [Background] Brody H. Medicine's ethical responsibility for health care reform--the Top Five list. N Engl J Med. 2010 Jan 28;362(4):283-5. doi: 10.1056/NEJMp0911423. Epub 2009 Dec 23. No abstract available. PMID 20032315
- [Background] Saslow D, Boetes C, Burke W, Harms S, Leach MO, Lehman CD, Morris E, Pisano E, Schnall M, Sener S, Smith RA, Warner E, Yaffe M, Andrews KS, Russell CA; American Cancer Society Breast Cancer Advisory Group. American Cancer Society guidelines for breast screening with MRI as an adjunct to mammography. CA Cancer J Clin. 2007 Mar-Apr;57(2):75-89. doi: 10.3322/canjclin.57.2.75. PMID 17392385
- [Background] Carlson RW, Allred DC, Anderson BO, Burstein HJ, Carter WB, Edge SB, Erban JK, Farrar WB, Forero A, Giordano SH, Goldstein LJ, Gradishar WJ, Hayes DF, Hudis CA, Ljung BM, Mankoff DA, Marcom PK, Mayer IA, McCormick B, Pierce LJ, Reed EC, Sachdev J, Smith ML, Somlo G, Ward JH, Wolff AC, Zellars R; National Comprehensive Cancer Network. Invasive breast cancer. J Natl Compr Canc Netw. 2011 Feb;9(2):136-222. doi: 10.6004/jnccn.2011.0016. No abstract available. PMID 21310842
- [Background] Khatcheressian JL, Wolff AC, Smith TJ, Grunfeld E, Muss HB, Vogel VG, Halberg F, Somerfield MR, Davidson NE; American Society of Clinical Oncology. American Society of Clinical Oncology 2006 update of the breast cancer follow-up and management guidelines in the adjuvant setting. J Clin Oncol. 2006 Nov 1;24(31):5091-7. doi: 10.1200/JCO.2006.08.8575. Epub 2006 Oct 10. PMID 17033037
- [Background] Harris L, Fritsche H, Mennel R, Norton L, Ravdin P, Taube S, Somerfield MR, Hayes DF, Bast RC Jr; American Society of Clinical Oncology. American Society of Clinical Oncology 2007 update of recommendations for the use of tumor markers in breast cancer. J Clin Oncol. 2007 Nov 20;25(33):5287-312. doi: 10.1200/JCO.2007.14.2364. Epub 2007 Oct 22. PMID 17954709
- [Background] Rojas MP, Telaro E, Russo A, Moschetti I, Coe L, Fossati R, Palli D, del Roselli TM, Liberati A. Follow-up strategies for women treated for early breast cancer. Cochrane Database Syst Rev. 2005 Jan 25;(1):CD001768. doi: 10.1002/14651858.CD001768.pub2. PMID 15674884
- [Background] Khatcheressian JL, Hurley P, Bantug E, Esserman LJ, Grunfeld E, Halberg F, Hantel A, Henry NL, Muss HB, Smith TJ, Vogel VG, Wolff AC, Somerfield MR, Davidson NE; American Society of Clinical Oncology. Breast cancer follow-up and management after primary treatment: American Society of Clinical Oncology clinical practice guideline update. J Clin Oncol. 2013 Mar 1;31(7):961-5. doi: 10.1200/JCO.2012.45.9859. Epub 2012 Nov 5. PMID 23129741
- [Background] Dinan MA, Curtis LH, Hammill BG, Patz EF Jr, Abernethy AP, Shea AM, Schulman KA. Changes in the use and costs of diagnostic imaging among Medicare beneficiaries with cancer, 1999-2006. JAMA. 2010 Apr 28;303(16):1625-31. doi: 10.1001/jama.2010.460. PMID 20424253
- [Background] Breslin TM, Banerjee M, Gust C, Birkmeyer NJ. Trends in advanced imaging use for women undergoing breast cancer surgery. Cancer. 2013 Mar 15;119(6):1251-6. doi: 10.1002/cncr.27838. Epub 2012 Dec 4. PMID 23212691
- [Background] Lostumbo L, Carbine NE, Wallace J. Prophylactic mastectomy for the prevention of breast cancer. Cochrane Database Syst Rev. 2010 Nov 10;(11):CD002748. doi: 10.1002/14651858.CD002748.pub3. PMID 21069671
- [Background] Tuttle TM, Habermann EB, Grund EH, Morris TJ, Virnig BA. Increasing use of contralateral prophylactic mastectomy for breast cancer patients: a trend toward more aggressive surgical treatment. J Clin Oncol. 2007 Nov 20;25(33):5203-9. doi: 10.1200/JCO.2007.12.3141. Epub 2007 Oct 22. PMID 17954711
- [Background] Yao K, Winchester DJ, Czechura T, Huo D. Contralateral prophylactic mastectomy and survival: report from the National Cancer Data Base, 1998-2002. Breast Cancer Res Treat. 2013 Dec;142(3):465-76. doi: 10.1007/s10549-013-2745-1. Epub 2013 Nov 12. PMID 24218052
- [Background] Katz SJ, Morrow M. Contralateral prophylactic mastectomy for breast cancer: addressing peace of mind. JAMA. 2013 Aug 28;310(8):793-4. doi: 10.1001/jama.2013.101055. No abstract available. PMID 23907558
- [Background] Roohan PJ, Bickell NA, Baptiste MS, Therriault GD, Ferrara EP, Siu AL. Hospital volume differences and five-year survival from breast cancer. Am J Public Health. 1998 Mar;88(3):454-7. doi: 10.2105/ajph.88.3.454. PMID 9518982
- [Background] Nattinger AB, Laud PW, Bajorunaite R, Sparapani RA, Freeman JL. An algorithm for the use of Medicare claims data to identify women with incident breast cancer. Health Serv Res. 2004 Dec;39(6 Pt 1):1733-49. doi: 10.1111/j.1475-6773.2004.00315.x. PMID 15533184
- [Background] Charlson ME, Pompei P, Ales KL, MacKenzie CR. A new method of classifying prognostic comorbidity in longitudinal studies: development and validation. J Chronic Dis. 1987;40(5):373-83. doi: 10.1016/0021-9681(87)90171-8. PMID 3558716
- [Background] Elixhauser A, Steiner C, Harris DR, Coffey RM. Comorbidity measures for use with administrative data. Med Care. 1998 Jan;36(1):8-27. doi: 10.1097/00005650-199801000-00004. PMID 9431328
- See also: Choosing Wisely — http://www.choosingwisely.org
- See also: American Society of Breast Surgeons. Official statements. — https://www.breastsurgeons.org/new_layout/about/statements/